CLINICAL TRIAL: NCT02854592
Title: Intravenous Thrombolysis Registry for Chinese Ischemic Stroke Within 4.5 h Onset
Acronym: INTRECIS
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurology department, General Hospital of Shenyang Military Region
Other Study IDs: k2016-11
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke
Keywords: rtPA; urokinase
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator; Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rtPA: Intravenous rt-PA thrombolysis shall be administered within 4.5 h after symptom onset, at a dose of 0.9 mg/kg body weight (maximum, 90 mg), with 10% of the dose given as a bolus over 1 min and the remaining 90% infused over 60 min.
  Interventions: Drug: rtPA
- urokinase: 1,000,000-1,500,000 units of urokinase intravenous infused over 30 minutes within 4.5 h of stroke onset .
  Interventions: Drug: urokinase

INTERVENTIONS:
Drug: rtPA — intravenous thrombolysis with rtPa
  Other Names: alteplase
  Groups: rtPA
Drug: urokinase — intravenous thrombolysis with urokinase
  Groups: urokinase

SUMMARY:
Stroke is one of the leading causes of death and disability in China. Intravenous thrombolysis with recombinant tissue plasminogen activator (rtPA) improves the outcome for ischemic stroke patients who can be treated within 4.5 hours of symptom onset. In China, in addition to rt-PA, intravenous urokinase within 6 h has also been recommended by the 2010 Chinese Guidelines for the Diagnosis and Treatment of Patients with Acute Ischemic Stroke, and supported by evidence from two intravenous urokinase thrombolysis trials. Urokinase is used more frequently than rt-PA, mainly because it is cheaper. To describe Chinese experience with thrombolytic therapy for Ischemic Stroke within 4.5h onset, we designed a multicenter, prospective, registry study. The aim of INtravenous Thrombolysis REgistry for Chinese Ischemic Stroke within 4.5 h onset（INTRECIS）was to assess the safety and efficacy of intravenous rtPA, urokinase as thrombolytic therapy within the first 4.5 h of onset of acute ischaemic stroke.

DETAILED DESCRIPTION:
INTRECIS is a prospective multicenter registry using data from 60 centres in the North China. Consecutive patients with acute ischemic stroke who are treated with intravenous rtPA, urokinase within 4.5 hours of symptom onset in 60 centres of the North China will be eligible for this registry. Patient involvement in the registry shall not influence any treatment decision. Patients will undergo a complete diagnostic work up including a clinical neurological examination using the National Institutes of Health Stroke Scale (NIHSS) score, laboratory examination, brain and neurovascular imaging, echocardiography, 24-hours ECG. Clinical outcome will be evaluated on day 1 and day 14 using the National Institute of Health Stroke Scale (NIHSS) score, evaluated at 3 months using modified Rankin Scale score (mRS) and assessing adverse events. The proportion of patients with excellent outcome (mRS 0 to 1) at 3 months after treatment will serve as the primary outcome. Secondary outcome measures will include independent functional outcome (mRS 0 to 2), changes in NIHSS at 1 and 14 day compared with baseline, symptomatic intracerebral haemorrhage, recurrent stroke and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ischemic stroke diagnosed by CT or MRI
* first stroke onset or past stroke without obvious neurological deficit (mRS≤1)
* Time from onset to treatment: ≤ 4.5 hours
* Treatment with intravenous rtPA or urokinase
* Signed informed consent by patient self or legally authorized representatives

Exclusion Criteria:

* History of subarachnoid hemorrhage, intracranial hemorrhage and hemorrhagic cerebral infarction
* Obvious head injuries or strokes within 3 months
* Intracranial tumor, arteriovenous malformation or aneurysm
* Intracranial or spinal cord surgery within 3 months
* Gastrointestinal or urinary tract hemorrhage within the previous 21 days
* Blood glucose < 50 mg/dl (2.7mmol/L)
* Heparin therapy or oral anticoagulation therapy within 48 hours
* Oral warfarin is being taken and INR>1.6
* Severe systemic disease which is expected to survive less than 3 months
* Major surgery within 1 month
* Uncontrolled hypertension (>180/100 mmHg)
* Platelet count < 10×109／L
* Patients who have been involved in other clinical trials within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke within 4.5 hours of symptom onset
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Excellent outcome at 3 months | 90 days
  The proportion of patients with excellent outcome (modified Rankin Score 0 to 1) at 3 months after stroke onset

SECONDARY OUTCOMES:
Functional independence at 3 months after stroke onset | 90 days
  the proportion of patients with functional independence (modified Rankin Scale, mRS, score 0-2) at 3 months after stroke onset
Symptomatic intracerebral haemorrhage | 22-36 hours
  Symptomatic intracranial haemorrhages defined as NIHSS score increase ≥4 caused by intracranial hemorrhage
Recurrent stroke | 90 days
  New stroke or TIA within 3 months
All-cause mortality | 1 day, 14 days, 90 days
  Death from all-cause death, stroke events or cardiovascular events
changes in NIHSS score | 1 day, 14 days
  changes in NIHSS score at 1 day and 14 days, compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Sheng Chen, Study Director — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Wang Y, Wu D, Zhao X, Ma R, Guo X, Wang C, Liu L, Zhao W, Wang Y. Hospital resources for urokinase/recombinant tissue-type plasminogen activator therapy for acute stroke in Beijing. Surg Neurol. 2009 Aug;72 Suppl 1:S2-7. doi: 10.1016/j.surneu.2007.12.028. Epub 2008 Apr 18. PMID 18423545
- [Background] European Stroke Organisation (ESO) Executive Committee; ESO Writing Committee. Guidelines for management of ischaemic stroke and transient ischaemic attack 2008. Cerebrovasc Dis. 2008;25(5):457-507. doi: 10.1159/000131083. Epub 2008 May 6. PMID 18477843
- [Derived] Cui Y, Wang XH, Zhao Y, Chen SY, Sheng BY, Wang LH, Chen HS. Association of serum biomarkers with early neurologic improvement after intravenous thrombolysis in ischemic stroke. PLoS One. 2022 Oct 31;17(10):e0277020. doi: 10.1371/journal.pone.0277020. eCollection 2022. PMID 36315566
- [Derived] Cui Y, Yao ZG, Chen HS. Intravenous thrombolysis with 0.65 mg/kg r-tPA may be optimal for Chinese mild-to-moderate stroke. Front Neurol. 2022 Sep 20;13:989907. doi: 10.3389/fneur.2022.989907. eCollection 2022. PMID 36203975
- [Derived] Cui Y, Wang XH, Zhao Y, Chen SY, Sheng BY, Wang LH, Chen HS. Change of Serum Biomarkers to Post-Thrombolytic Symptomatic Intracranial Hemorrhage in Stroke. Front Neurol. 2022 Jun 2;13:889746. doi: 10.3389/fneur.2022.889746. eCollection 2022. PMID 35720096
- [Derived] Cui Y, Meng WH, Chen HS. Early neurological deterioration after intravenous thrombolysis of anterior vs posterior circulation stroke: a secondary analysis of INTRECIS. Sci Rep. 2022 Feb 24;12(1):3163. doi: 10.1038/s41598-022-07095-6. PMID 35210531
- [Derived] Wang X, Li X, Xu Y, Li R, Yang Q, Zhao Y, Wang F, Sheng B, Wang R, Chen S, Wang L, Shen L, Hou X, Cui Y, Wang D, Peng B, Anderson CS, Chen H; INTRECIS Investigators. Effectiveness of intravenous r-tPA versus UK for acute ischaemic stroke: a nationwide prospective Chinese registry study. Stroke Vasc Neurol. 2021 Dec;6(4):603-609. doi: 10.1136/svn-2020-000640. Epub 2021 Apr 26. PMID 33903179